CLINICAL TRIAL: NCT04500964
Title: Transcatheter Aortic Valve Replacement for Failed Transcatheter Aortic Valve. An International Registry
Brief Title: Transcatheter Aortic Valve Replacement for Failed Transcatheter Aortic Valve
Status: Completed | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Luca Testa, Interventional Cardiology, IRCCS Policlinico S. Donato
Other Study IDs: TRANSIT
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Failed Transcather Aortic Valve

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- failed transcather aortic valve (Stenotic)
  Interventions: Device: TAVR
- failed transcather aortic valve (Regurgitation)
  Interventions: Device: TAVR
- failed transcather aortic valve (Regurgitation and stenotic))
  Interventions: Device: TAVR

INTERVENTIONS:
Device: TAVR — Trancatheter aortic valve replacement

SUMMARY:
Patients with failed transcather aortic valve (stenotic, regurgitant, both) and indication to further transcatheter aortic valve replacement (TAVR).

The purpouse of this study is to evaluate the indication to a second TAVR, the selection criteria of the second transcatheter aortic valve, procedural and clinical outcomes.

The primary endpoint of the study is overall mortality and Cardiovascular mortality at 1 year

ELIGIBILITY:
Inclusion Criteria:

* Patients with failed transcather aortic valve (stenotic, regurgitant, both) and indication to further transcatheter aortic valve replacement (TAVR).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with failed transcather aortic valve
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 1 year
  Overall mortality and Cardiovascular mortality at 1 year

SECONDARY OUTCOMES:
VARC-3 Events | 1 year
  Cerebrovascular events, bleeding complications, periprocedural MI, conduction disturbances, BVF, procedural success, device success, AKI (all according to VARC-2).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Testa L, Casenghi M, Criscione E, Van Mieghem NM, Tchetche D, Asgar AW, De Backer O, Latib A, Reimers B, Stefanini G, Trani C, Giannini F, Bartorelli A, Wojakowski W, Dabrowski M, Jagielak D, Banning AP, Kharbanda R, Moreno R, Schofer J, Brinkmann C, van Royen N, Pinto D, Serra A, Segev A, Giordano A, Brambilla N, Agnifili M, Rubbio AP, Squillace M, Oreglia J, Tanja R, McCabe JM, Abizaid A, Voskuil M, Teles R, Zoccai GB, Sondergaard L, Bedogni F. Prosthesis-patient mismatch following transcatheter aortic valve replacement for degenerated transcatheter aortic valves: the TRANSIT-PPM international project. Front Cardiovasc Med. 2022 Jul 29;9:931207. doi: 10.3389/fcvm.2022.931207. eCollection 2022. PMID 35966561
- [Derived] Testa L, Agnifili M, Van Mieghem NM, Tchetche D, Asgar AW, De Backer O, Latib A, Reimers B, Stefanini G, Trani C, Colombo A, Giannini F, Bartorelli A, Wojakowski W, Dabrowski M, Jagielak D, Banning AP, Kharbanda R, Moreno R, Schofer J, van Royen N, Pinto D, Serra A, Segev A, Giordano A, Brambilla N, Popolo Rubbio A, Casenghi M, Oreglia J, De Marco F, Tanja R, McCabe JM, Abizaid A, Voskuil M, Teles R, Biondi Zoccai G, Bianchi G, Sondergaard L, Bedogni F. Transcatheter Aortic Valve Replacement for Degenerated Transcatheter Aortic Valves: The TRANSIT International Project. Circ Cardiovasc Interv. 2021 Jun;14(6):e010440. doi: 10.1161/CIRCINTERVENTIONS.120.010440. Epub 2021 Jun 7. PMID 34092097